CLINICAL TRIAL: NCT01962766
Title: Myofunctionnal Therapy on Nasal Breathing and Orthodontic Corrections Stability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Nelly Huynh, Assistant research professor, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NH-13-OP-DegluLang; 13-104-CERES-P (Other: UMontreal - CERES)
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Mouth Breathing; Atypic Swallowing; Low Resting Position of Tongue
MeSH Terms: conditions — Mouth Breathing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- complete myofunctionnal therapy (Active Comparator): complete therapy (at least 5 sessions) to correct their swallowing pattern and tongue position
  Interventions: Behavioral: Myofunctionnal therapy
- instructions (Experimental): instructions to modify their tongue position (1 session)
  Interventions: Behavioral: instructions

INTERVENTIONS:
Behavioral: Myofunctionnal therapy
  Arms: complete myofunctionnal therapy
Behavioral: instructions
  Arms: instructions

SUMMARY:
The current research project aims to study the efficacy of myofunctional therapy and its orthodontic long-term outcomes.

DETAILED DESCRIPTION:
The current research project aims to study the efficacy of myofunctional therapy and its orthodontic long-term outcomes, such as: 1) Is treating a low tongue position and lip closure at rest sufficient for orthodontic short and long-term outcomes? 2) Does treating atypical swallowing along with an incorrect tongue position help achieve and maintain higher outcomes of the myofucntional and orthodontic treatments?

ELIGIBILITY:
Inclusion Criteria:

* Between 6 and 14 years old
* Atypical or immature swallowing pattern and lower position of the tongue at rest
* Be an orthodontic patient treated at the Faculty of Dentistry, Université de Montreal
* Speak and understand French without assistance
* Be in good health (without neurological or psychiatric syndrome)
* Agree to participate and sign the consent form research

Exclusion Criteria:

* Non compliance to clinical visits (eg too many missed visits)
* Patients who had previous orthodontic treatments
* Syndrome or known systemic disease (chronic cardiopulmonary or neuromuscular disease, dysmorphia, major craniofacial abnormalities)

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
respiration mode | 6 months following therapy
  orthophonist speech assessment, including nasal or mouth respiration, swallowing pattern and tongue resting position

SECONDARY OUTCOMES:
tongue resting position | 6 months following therapy
  orthophonist speech assessment, including nasal or mouth respiration, swallowing pattern and tongue resting position

OTHER OUTCOMES:
swallowing pattern | 6 months following therapy
  orthophonist speech assessment, including nasal or mouth respiration, swallowing pattern and tongue resting position

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique d'orthodontie - Université de Montréal, Montreal, Quebec, Canada